CLINICAL TRIAL: NCT03648892
Title: Brain Dopamine Function in Human Obesity
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 180132; 18-DK-0132
Record Dates: First submitted 2018-08-24; First posted 2018-08-28 (Actual); Results first posted 2023-05-03 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2022-05

CONDITIONS: Obesity; Healthy Volunteers; Overweight
Keywords: Dopamine Response; Energy Expenditure; Neurocognitive Function; Obesity
MeSH Terms: conditions — Obesity; Overweight | interventions — Raclopride; N-((1-allyl-2-pyrrolidinyl)methyl)-5-(3-fluoropropyl)-2,3-dimethoxybenzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Main (Other): Healthy volunteers, within three BMI strata, under controlled overnight fasting conditions following a period of dietary stabilization
  Interventions: Drug: [c11] raclopride; Drug: [18F]fallypride

INTERVENTIONS:
Drug: [c11] raclopride — The present study will attempt to resolve the controversy by measuring D2BP using both [18F]fallypride and [11C]raclopride in 39 adults, 13 within each of three BMI strata to represent a large BMI range, under controlled overnight fasting conditions following a period of dietary stabilization. The primary aims are to estimate the mathematical relationship between striatal D2BP and BMI and determine the within-subject correlations of D2BP derived from [18F]fallypride and [11C]raclopride.
Drug: [18F]fallypride — The present study will attempt to resolve the controversy by measuring D2BP using both [18F]fallypride and [11C]raclopride in 39 adults, 13 within each of three BMI strata to represent a large BMI range, under controlled overnight fasting conditions following a period of dietary stabilization. The primary aims are to estimate the mathematical relationship between striatal D2BP and BMI and determine the within-subject correlations of D2BP derived from [18F]fallypride and [11C]raclopride.

SUMMARY:
Background:

Dopamine is a natural chemical in the brain that may influence eating behavior and physical activity. Researchers want to measure the brain s dopamine activity and understand how it differs in people with obesity.

Objective:

To better understand how brain function, particularly dopamine activity, relates to body weight and eating behavior.

Individuals may be able to participate if they:

Have a BMI of at least 18.5 kg/m2

Are weight-stable and generally healthy

Are between ages 18-45 years

Have normal blood pressure

Are not using illegal drugs (based on urine drug screen)

Are not following a special diet

Do not have metal implants

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Questionnaires and an interview to see if it is safe to have a PET/MRI scan
* Fasting blood and urine tests
* Participants will eat a special diet given to them for the 5 days before their inpatient visit.

Participants will have a 5-day inpatient visit. Some days include blood and urine tests. Each day includes surveys and tests to measure habits and likes/dis-likes. A sample schedule may be:

Day 1: Participants will wear a monitor that uses a needle below the skin to measure glucose. Their body fat will be measured with low-dose x-rays

Day 2: Participants will have a PET scan. They will lie on a table that slides in and out of a donut-shaped scanner. They will be injected with a small amount of a radioactive substance and wear a cap on their head.

Day 3: Participants will have an MRI. They will lie on a table that slides in and out of a scanner.

Day 4: Participants will have another PET scan. This time, they will drink a milk shake during a break from the scanner. Then, they will go back inside the scanner for the end of their scan.

Day 5: Participants will wear a hood for up to 40 minutes to measure their breathing. They will also drink special water and collect samples of their urine to measure the rate they burn energy.

For 12 months after the visit, participants will track their weight and physical activity daily using a special scale and activity monitor. A few times over the year, the study team will send participants special activity monitors to use for 7 days at a time.

Participants will have an in-person 1-day follow-up visit. This includes most tests except for PET scanning....

DETAILED DESCRIPTION:
Evidence from neuroimaging studies indicates that aberrant functionality in brain regions that support reward processing and habit formation may be related to an individual's eating behavior and obesity propensity. In particular, our previous research found that increased dopamine D2 receptor binding potential (D2BP) in the dorsal and lateral striatum was positively related to opportunistic eating behaviors, body fat, and body mass index (BMI). However, our findings were contrary to highly-cited previous reports of D2BP correlating with BMI in the opposite direction. The primary aim of this study is to elucidate the reasons for the conflicting results that used somewhat different methodologies. Specifically, our previous study used positron emission tomography (PET) to measure D2BP using the dopamine D2 receptor antagonist radioligand [18F]fallypride following a period of dietary stabilization and 3 hours after a standardized breakfast. Reports finding correlations between D2BP and BMI in the opposite direction have typically investigated subjects with higher BMI using the D2 receptor antagonist radioligand [11C]raclopride. Furthermore, previous studies were typically conducted in the fasted state, but the subjects' prior food intake was not well-controlled. The present study will attempt to resolve the controversy by measuring D2BP using both [18F]fallypride and [11C]raclopride in 39 adults, 13 within each of three BMI strata to represent a large BMI range, under controlled overnight fasting conditions following a period of dietary stabilization. The primary aims are to estimate the mathematical relationship between striatal D2BP and BMI and determine the within-subject correlations of D2BP derived from [18F]fallypride and [11C]raclopride.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18-45 years, male and female
* Consent to undergoing PET scanning
* Body mass index (BMI) greater than or equal to 18.5 kg/m^2
* Weight stable (less than plus or minus 5% change in the past month)
* Written informed consent
* Estimated intelligence quotient (IQ) greater than or equal to 70, as determined by the National Adult Reading Test (NART) (Scores below 70 are indicative of mental retardation; IQ has been related to alterations in brain structure and function that may confound neuroimaging measures. Failure to meet this eligibility criteria will be documented in the record and communicated to the potential participant as ineligibility based on reading test results )

EXCLUSION CRITERIA:

* Age 46 or greater (Age is a significant confound in the relationship between BMI and dopamine. Dopamine binding has been shown to drastically decrease in the fifth decade of life.
* Body weight > 400 lbs. (weight limit of PET scanner)
* Weigh less than 80% of maximum lifetime weight
* BMI < 18.5 kg/m2
* Past or present history of neurological or psychiatric disease (e.g., depression, anxiety, substance use disorder or psychosis), or eating disorders (e.g., anorexia nervosa, bulimia nervosa, or binge eating disorder) as determined by research team upon review of history/physical, Eating Disorder Examination-Questionnaire and Self-Rated Level 1 Cross-Cutting Symptom Measure.
* Blood pressure >140/90 mm Hg
* Evidence/history of cancer, metabolic disease (e.g. thyroid disease, diabetes) or cardiovascular disease (e.g. coronary artery disease, myocardial infarction, stroke, atherosclerosis), or disease that may influence metabolism
* Current use of prescription medication or other drug that may influence metabolism (diet/weight-loss medication, asthma medication, psychiatric medications such as antidepressants, anti-anxiety medications, and stimulants for attention-deficit/hyperactivity disorder (ADHD), corticosteroids or other medications at the discretion of the PI and/or study team)
* Pregnancy, lactation at any time during study/follow-up period (women only)
* Evidence of vigorous exercising in order to lose weight, change body shape, or to counteract the effects of eating
* Previous bariatric surgery
* Evidence of nicotine dependence as determined by Fagerstrom score greater than or equal to 3 (including chewing or smoking tobacco), any drug use (amphetamines, cocaine, heroin, marijuana), or problematic alcohol use (i.e. diagnosis of alcohol use disorder: meeting greater than or equal to 2 of 11 criteria in past 12 months, ranging from drinking more/longer than intended to experiencing withdrawal symptoms); report of binge drinking: greater than or equal to 5 drinks in 2 hours or greater than or equal 4 drinks in

  2 hours for men and women, respectively) over the previous 6 months.
* Volunteers with strict dietary concerns (e.g. kosher diet, milk allergy or lactose intolerance, or food allergies)
* Caffeine consumption > 300 mg/day (roughly greater than or equal to 3 cups coffee or 2-3 energy drinks)
* Having metal implants incompatible with MRI (for example, pacemakers, metallic prostheses such as cochlear implants or heart valves, shrapnel fragments, etc.).
* Having had previous radiation exposure within the last year for either medical or research purposes (e.g. X-rays, PET scans, etc.) that would exceed research limits. Excessive radiation exposure will be determined at the discretion of the PI and/or study team
* Are claustrophobic to a degree that they would feel uncomfortable in the MRI machine.
* Non-English speakers.
* Cannot commit to the schedule of visits to the Clinical Research Center as required by the study timeline

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2023-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Hall, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Darcey VL, Guo J, Chi M, Chung ST, Courville AB, Gallagher I, Herscovitch P, Howard R, La Noire M, Milley L, Schick A, Stagliano M, Turner S, Urbanski N, Yang S, Yim E, Zhai N, Zhou MS, Hall KD. Striatal dopamine tone is positively associated with adiposity in humans as determined by PET using dual dopamine type-2 receptor antagonist tracers. Mol Psychiatry. 2025 Aug;30(8):3708-3717. doi: 10.1038/s41380-025-02960-y. Epub 2025 Apr 6. PMID 40188315
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-DK-0132.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Dopamine D2/3 Receptor Antagonists: Healthy volunteers, within three Body Mass Index (BMI) strata, under controlled overnight fasting conditions following a period of dietary stabilization. The present study will attempt to resolve the controversy surrounding the relationship between BMI and dopamine D2 receptor availability by measuring D2 Receptor Binding Potential (D2BP) using both [18F]Fallypride and [11C]Raclopride in pseudorandom order during days 2-5 of the inpatient stay.
Period: Overall Study
Arm/Group | Dopamine D2/3 Receptor Antagonists
Started | 61
Completed | 61
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dopamine D2/3 Receptor Antagonists
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.67 (7.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 32
  White | 18
  More than one race | 1
  Unknown or Not Reported | 3
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.09 (8.21)

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Striatal D2 Receptor Binding Potential (D2BP) as Measured by [18F]Fallypride and [11C]Raclopride Time-activity Curves
Description: Correlations between striatal D2BP via [18F]Fallypride and striatal D2BP via [11C]Raclopride is obtained.
  Pearson's correlation coefficient is used with a possible range between -1 to 1 indicating strong association in the same direction as correlation is closer to 1, strong association in opposite direction as correlation is closer to -1, and no association as correlation is closer to 0.
Time Frame: assessed at Days 2-5
Population: Only 54 participants completed striatal D2 Receptor Binding Potential (D2BP) as measured by [18F]Fallypride and [11C]Raclopride.
Measure: Number (95% Confidence Interval); unit: Correlation Coefficient
Arm/Group | Dopamine D2/3 Receptor Antagonists
Number analyzed (Participants) | 54
Correlation Coefficient | 0.468 [.229 to .654]

2. Primary Outcome: Relationship Between Striatal D2BP and BMI is Quadratic or Linear
Description: Coefficient estimate of the quadratic term of BMI in quadratic regression is obtained and Coefficient estimate of the linear term of BMI in simple linear regression is obtained.
Time Frame: assessed at Days 2-5
Population: Only 57 participants had non-missing values of D2BP via [18F]Fallypride and 56 participants had non-missing values of D2BP via 11C]Raclopride. Thus, the total number of participants analyzed is different for each of rows below.
Measure: Number (95% Confidence Interval); unit: Coefficient estimate
Arm/Group | Dopamine D2/3 Receptor Antagonists
Number analyzed (Participants) | 61
Coefficient estimate
  Coefficeint of quadratic determination with D2BP Via [18F]Fallypride: number analyzed (Participants) | 57
  Coefficeint of quadratic determination with D2BP Via [18F]Fallypride | -0.022 [-0.047 to 0.003]
  Coefficient of quadratic determination with D2BP Via [11C]Raclopride: number analyzed (Participants) | 56
  Coefficient of quadratic determination with D2BP Via [11C]Raclopride | -0.001 [-0.003 to 0.001]
  Coefficient of linear determination with D2BP Via [18F]Fallypride: number analyzed (Participants) | 57
  Coefficient of linear determination with D2BP Via [18F]Fallypride | -0.032 [-0.186 to 0.121]
  Coefficient of linear determination with D2BP Via [11C]Raclopride: number analyzed (Participants) | 56
  Coefficient of linear determination with D2BP Via [11C]Raclopride | -0.027 [-0.039 to -0.015]

3. Primary Outcome: Change in Striatal Dopamine D2BP After a Palatable Meal
Description: To determine the effect of palatable meal consumption on striatal D2BP using [11C]Raclopride
Time Frame: assessed at Days 2-5
Population: Only 50 participants had non-missing values of change in striatal dopamine D2BP after a palatable meal.
Measure: Mean (Standard Deviation); unit: Binding Potential
Arm/Group | Dopamine D2/3 Receptor Antagonists
Number analyzed (Participants) | 50
Binding Potential | -0.0164 (0.23)

4. Primary Outcome: Correlation Between Change in Striatal Dopamine D2BP After a Palatable Meal and BMI
Description: To determine association between change in striatal dopamine D2BP after a palatable meal consumption and BMI. Binding potential estimates will be estimated within subjects using [11C]Raclopride
Time Frame: assessed at Days 2-5
Population: Only 50 participants had non-missing values of both change in striatal dopamine D2BP after palatable meal.
Measure: Number (95% Confidence Interval); unit: Correlation Coefficient
Arm/Group | Dopamine D2/3 Receptor Antagonists
Number analyzed (Participants) | 50
Correlation Coefficient | 0.276 [-0.002 to 0.515]

5. Secondary Outcome: Associations Between Behavioral Performance on Food Go/No Go Computer Task and Striatal D2BP
Description: Exploratory analyses of correlations between behavioral performance on Food Go/No Go computer task measured by No Go accuracy as commission errors and striatal D2BP via [18F]Fallypride and via [11C]Raclopride.
  Pearson's correlation coefficient is used with a possible range between -1 to 1 indicating strong association in the same direction as correlation is closer to 1, strong association in opposite direction as correlation is closer to -1, and no association as correlation is closer to 0.
Time Frame: assessed at Days 2-5
Population: Only 54 participants had non-missing values of behavioral performance and striatal D2BP via [18F]Fallypride and 53 participants had non-missing values of behavioral performance and striatal D2BP via 11C]Raclopride. Thus, the total number of participants analyzed is different for each of rows below.
Measure: Number (95% Confidence Interval); unit: Correlation Coefficient
Arm/Group | Dopamine D2/3 Receptor Antagonists
Number analyzed (Participants) | 61
Correlation Coefficient
  D2BP Via [18F]Fallypride: number analyzed (Participants) | 54
  D2BP Via [18F]Fallypride | 0.156 [-0.116 to 0.407]
  D2BP Via [11C]Raclopride: number analyzed (Participants) | 53
  D2BP Via [11C]Raclopride | 0.047 [-0.226 to 0.313]

6. Secondary Outcome: Associations Between ad Libitum Meal Consumption and Striatal D2 Receptor (D2R)
Description: Exploratory analyses of correlations between eating behavior measured by ad libitum food intake at a single meal and striatal D2R via [18F]Fallypride and via [11C]Raclopride
Time Frame: assessed at Days 2-5
Population: Only 53 participants had non-missing values of ad libitum meal consumption and striatal D2R via [18F]Fallypride and 52 participants had non-missing values of ad libitum meal consumption and striatal D2R via [11C]Raclopride. Thus, the total number of participants analyzed is different for each of rows below.
Measure: Number (95% Confidence Interval); unit: Correlation Coefficient
Arm/Group | Dopamine D2/3 Receptor Antagonists
Number analyzed (Participants) | 61
Correlation Coefficient
  D2R Via [18F]Fallypride: number analyzed (Participants) | 53
  D2R Via [18F]Fallypride | -0.037 [-0.305 to 0.235]
  D2R Via [11C]Raclopride: number analyzed (Participants) | 52
  D2R Via [11C]Raclopride | -0.118 [-0.379 to 0.160]

7. Secondary Outcome: Associations Between Brain Metabolite GABA Via MRS and Striatal D2BP Via [18F]Fallypride
Description: Exploratory analyses of correlations between brain metabolite GABA via magnetic resonance spectroscopy (MRS) and striatal D2BP via [18F]Fallypride.
  Pearson's correlation coefficient is used with a possible range between -1 to 1 indicating strong association in the same direction as correlation is closer to 1, strong association in opposite direction as correlation is closer to -1, and no association as correlation is closer to 0.
Time Frame: assessed at Days 2-5
Population: Only 33 participants had non-missing values of brain metabolite gamma-aminobutyric acid (GABA) via MRS and striatal D2BP via [18F]Fallypride. Thus, the total number of participants analyzed is different for each of rows below.
Measure: Number (95% Confidence Interval); unit: Correlation Coefficiant
Arm/Group | Dopamine D2/3 Receptor Antagonists
Number analyzed (Participants) | 33
Correlation Coefficiant | -0.254 [-0.549 to 0.098]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Dopamine D2/3 Receptor Antagonists
All-Cause Mortality (participants affected / at risk) | 0/61
Serious Adverse Events (participants affected / at risk) | 0/61
Other Adverse Events (participants affected / at risk) | 3/61
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dopamine D2/3 Receptor Antagonists (N=61)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/92/NCT03648892/Prot_SAP_000.pdf